CLINICAL TRIAL: NCT03508518
Title: Improving Access to Psychiatric Care and the Fluidity of Care Pathways for Patients Suffering From Mental Disorders in Primary Care in France: Evaluation of a Psychiatric Consultation-liaison System
Brief Title: Improving Access to Psychiatric Care for Patients in Primary Care
Acronym: DSPP-PSY
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: recruitment difficulties
Sponsor: University Hospital, Toulouse (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: RC31/17/0357; 2017-A03127-46 (Other: ID-RCB)
Record Dates: First submitted 2018-04-16; First posted 2018-04-25 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Mental Disorder
Keywords: Accessibility of health services; Access to psychiatric care; Consultation-liaison; General practitioner and psychiatrist collaboration; Care pathway
MeSH Terms: conditions — Mental Disorders | interventions — Psychiatry; dentin sialophosphoprotein

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Shared care device in psychiatry (DSPP) (Experimental): System focused on collaboration between general medicine (GP) and psychiatry, offering psychiatric assessment consultations and guidance for patient addressed by his/her GP. Referrals are made to the GP with support for care or the patient can be oriented to routine psychiatric care.
  Interventions: Other: Shared care device in psychiatry (DSPP)
- Care as usual (Active Comparator): Patient will have usual care :
  Psychiatric care available in the Haute Garonne: psychiatric consultation by a liberal psychiatrist or by a psychiatrist working in public health center
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: Shared care device in psychiatry (DSPP) — The GPs of the intervention group will be able to refer their patients to the DSPP or to the routine care. The patient has a nursing telephone interview prior to one or few more psychiatric consultations. The time to obtain the psychiatric consultation is measured into the 2 groups. In both groups, questionnaires will be sent to the patient and their medico-administrative data will be collected passively over a period of 6 months after inclusion
  Arms: Shared care device in psychiatry (DSPP)
Other: Usual Care — psychiatric care available in the Haute Garonne: psychiatric consultation by a liberal psychiatrist or by a psychiatrist working in public health center.
  Arms: Care as usual

SUMMARY:
Getting a consultation with a psychiatrist within an appropriate time is one of the main issues reported by general practitioners (GP) for patients suffering from mental disorders in primary care. Consultation liaison in psychiatry is a system focused on general medicine-psychiatry collaboration. The aim of the present study is to evaluate the impact of the consultation-liaison on the adequacy of the access time to a psychiatric consultation according to the degree of urgency evaluated by the GP.

DETAILED DESCRIPTION:
Faced with the saturation of the psychiatric care system, who recognizes the key role of the GP in mental health. Three-quarters of prescriptions for antidepressants and anxiolytics are performed by GPs, but less than one in four people with depression have been diagnosed and treated appropriately. The GPs describe difficulties in accessing psychiatric professionals and in particular to obtain a quick consultation with a psychiatrist. In different countries, psychiatric consultation-liaison (CL), centered on the collaboration of general medicine and psychiatry, have emerged. Two meta-analyzes and a Cochrane review were conducted on CL but no clinical trials were conducted in France. CL seems to improve patients' health at 3 months as well as their satisfaction and adherence to care. Results regarding the improvement of prescriptions from GP are encouraging. Better clinical trials are being requested and a need for medico-economic studies is also identified.

In France, a psychiatry CL was born in Toulouse in 2017, the "DSPP". The present study plans a 2 groups randomized clinical trial, one group of GPs having access to DSPP, the other not. For a period of 3 months, the GPs propose to any patient, for whom they want a psychiatric consultation, to participate in the study and address him/her to a psychiatrist. The DSPP is an evaluation center without long-term patient follow-up. Only patient referred by his/her GP can get into the DSPP.

ELIGIBILITY:
Inclusion Criteria:

* 15 years patient or older:
* presenting mental suffering or a frequent or severe mental disorder
* having consulted his GP who ask for psychiatric consultation
* having given its consent for the use of its medico-administrative data
* affiliated with the general health insurance scheme
* of which the GP is from Haute Garonne and is voluntary to participate in the study
* Free, informed and written consent signed by the participant and the investigator (at the latest on the day of inclusion and before any examination required by the research) and by one of the parents for minor participants

Exclusion Criteria:

* Patient with ongoing psychiatric follow-up
* Patient unable to answer questionnaires (unable to read or write)
* Patients receiving a measure of legal protection

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2018-08-28 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
Number of patients who had access to a consultation with a psychiatrist | 2 to 21 working days after inclusion
  Number of patients who had access to a consultation with a psychiatrist within 2 working days following the GP consultation for patients whose GP wishes an "urgent" consultation, within 7 working days for a "quick" consultation and within 21 working days for a "non-urgent" consultation.

SECONDARY OUTCOMES:
Number of days between M0 (GP consultation) and M1 (psychiatric consultation) | 6 months
  Number of days between M0 (GP consultation) and M1 (psychiatric consultation) collected passively on the bases of Health Insurance, Information Systems Medicalization Program (PMSI) and DSPP
Number of passages to psychiatric emergencies | 6 months
  Number of passages to psychiatric emergencies within 6 months M0 passively collected on the basis of the PMSI (Information Systems Medicalization Program) of psychiatric emergencies
Number of suicide attempts | 6 months
  Number of suicide attempts and suicides within 6 months following M0 passively collected on the basis of the PMSI of the psychiatric emergencies and the Health Insurance
Mental health status by Symptom Checklist (SCL) | date of inclusion, 1 month and 6 months after inclusion
  Mental health status measured at M0, 1 month and 6 months by questionnaires hand-delivered by the GP at M0 and sent at 1 and 6 months :
  - SCL-90-R scale: Scale exploring 9 symptomatic dimensions (somatization, obsession-compulsion, sensory traits, depression, anxiety, hostility, phobic anxiety, paranoid ideals, psychotic traits) by Likert scale in 5 points. Passing 15min.
Mental health status by Patient Health Questionnaire (PHQ) | date of inclusion, 1 month and 6 months after inclusion
  Mental health status measured at M0, 1 month and 6 months by questionnaires hand-delivered by the GP at M0 and sent at 1 and 6 months :
  - the PHQ-9 scale for the diagnosis of major depressive episode and the intensity of depression. 9 questions are rated from 0 to 3 by the patient, ie a score of severity ranging from 0 to 27.
Duration of prescription of different drugs | date of inclusion, 1 month and 6 months after inclusion
  Duration of prescription of a benzodiazepine, antidepressant, hypnotic and antipsychotic treatment passively collected on the bases of Health Insurance
Evaluation of compliance with antidepressant prescriptions | date of inclusion, 1 month and 6 months after inclusion
  Composite criterion for the evaluation of compliance with antidepressant prescriptions including drug type (first-line serotonin reuptake inhibitors (IRS): 0 or 1) and duration (6 months minimum: 0 or 1) with a total score of 0 to 2
Number of prescription treatment of mental disorders | date of inclusion, 1 month and 6 months after inclusion
  Number of prescription of a benzodiazepine, antidepressant, hypnotic and antipsychotic treatment passively collected on the bases of Health Insurance
Employment status | 6 months
  Occupation, without profession (Number and duration of sick leave within 6 months following M0, passively collected on the bases of Health Insurance)
Patient satisfaction | 1 month
  Patient satisfaction measured at 1 month of M0 by the Client Satisfaction Questionnaire (CSQ-8 scale)
Quality of life with EuroQol scale | 6 months
  Quality of life measured by the EuroQol (EQ-5D-5L) scale at M0 and 6 months by a clinical researcher by phone The EQ-5D-5L scale consists of 2 pages, a descriptive system EQ-5D and a visual analogue scale EQ . The descriptive system explores the following five dimensions: mobility, autonomy, usual activities, pain / discomfort and anxiety / depression. Each dimension is rated in 5 levels . The visual analogue scale is a vertical scale where the endpoints are labeled "best health imaginable" and "worst health imaginable"
GP satisfaction | 6 months
  GP satisfaction measured by questionnaire
Incremental Cost-Utility | 6 months
  to determine Incremental Cost-Utility collected passively on the bases of Health Insurance, PMSI and DSPP
Cost-Effectiveness Ratios of Patient Management Strategies | 6 months
  to determine Cost-Effectiveness Ratios of Patient Management Strategies collected passively by data on the bases of Health Insurance, PMSI and DSPP
Production costs | 6 months
  to determine production costs collected passively on the bases of Health Insurance, PMSI and DSPP

CONTACTS AND LOCATIONS:
Overall Officials: Sophie Prébois, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- University Hospital Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No